CLINICAL TRIAL: NCT02046551
Title: Atomoxetine's Effects On Nicotine Response And Stress Response In Smokers
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: funding lost
Sponsor: Yale University (Other)
Collaborators: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1305012021
Record Dates: First submitted 2014-01-23; First posted 2014-01-27 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Nicotine Dependence
Keywords: nicotine; smoking; atomoxetine; stress
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo
- Atomoxetine (Experimental): atomoxetine (40 mg/day)
  Interventions: Drug: Atomoxetine

INTERVENTIONS:
Drug: Atomoxetine
  Other Names: Strattera
  Arms: Atomoxetine
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate atomoxetine's effects on the rewarding and reinforcing effects of nicotine in a controlled human laboratory study with 24 otherwise healthy nicotine dependent subjects. It is hypothesized that atomoxetine will attenuate the negative effects of nicotine.

ELIGIBILITY:
Inclusion Criteria:

* female and male smokers, not treatment seeking, aged 18 to 55 years;
* history of smoking daily for the past 12 months, at least 5 cigarettes daily;
* CO level > 10ppm;
* for women: not pregnant as determined by pregnancy screening, nor breast feeding, and using acceptable birth control methods.

Exclusion Criteria:

* history of major medical illnesses including asthma or chronic obstructive lung disease, history or current gastrointestinal ulcer, hepatic or renal impairment, coronary artery disease, cardiac rhythm disturbances or other medical conditions that the study physician deems contraindicated for the subject to be in the study;
* regular use of psychotropic medication (antidepressants, antipsychotics, or anxiolytics)
* recent psychiatric diagnosis and treatment for Axis I disorders including major depression, bipolar affective disorder, schizophrenia and panic disorder within the past year. We will make an exception for the following Axis I diagnoses: nicotine dependence and alcohol or other drug dependence (i.e., cocaine, opioid) as long as they are not meeting abuse or dependence criteria within the past 3 months for alcohol or drug use;
* use of drugs that slow heart rate (eg, beta-blockers), which may increase the risk of bradycardia and AV block, or NSAIDs, which may increase potential for developing ulcers/active or occult gastrointestinal bleeding;
* known allergy to atomoxetine

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Nicotine Effects Questionnaire | Day 5
  Subjects will rate 6 items that are related to nicotine effect on a 100 mm scale, "not at all" to "extremely." The items are feeling the drug strength, feel "good" drug effects, feel "bad" drug effects, feel jittery, feel stimulated, and head rush. This instrument is an abbreviated version of a visual analog scale (VAS) and allows rapid detection of nicotine effects.
Nicotine Effects Questionnaire | Day 17
  Subjects will rate 6 items that are related to nicotine effect on a 100 mm scale, "not at all" to "extremely." The items are feeling the drug strength, feel "good" drug effects, feel "bad" drug effects, feel jittery, feel stimulated, and head rush. This instrument is an abbreviated version of a visual analog scale (VAS) and allows rapid detection of nicotine effects.

SECONDARY OUTCOMES:
Center for Epidemiologic Studies Depression (CES-D) scale | Day 5
  The Center for Epidemiologic Studies Depression (CES-D) scale is a 20-item self-report measure of depressive symptoms. The range of scores is from 0 to 60, with higher scores reflecting increased depressive symptoms 41. The CES-D does not heavily depend on pathological items compared with other scales such as the Beck Depression Inventory and does not define clinical depression.
Positive and Negative Affect Schedule (PANAS ) | Day 5
  Positive and Negative Affect Schedule (PANAS ) is a 20-item scale that assesses both negative and positive affective states. Subjects rate adjectives describing affective states on a scale of 1 to 5 using a specified time period (e.g., now, today, past week etc.). Scores are then added up to generate negative and positive scale scores.
The Profile of Mood States (POMS) | Day 5
  The Profile of Mood States (POMS) is a 72-item questionnaire which consists of adjectives commonly used to describe momentary mood states. It has been found to be sensitive to the mood-altering effects of drugs including nicotine. POMS has a 5-point objective rating scale (0=not at all to 5=extremely). There are eight mood states that this scale measures: (1) Anger, (2) Anxiety, (3) Confusion, (4) Depression, (5) Elation, (6) Fatigue, (7) Friendliness and (8) Vigor. POMS will be used during each session to measure effects of atomoxetine or nicotine on mood.
Center for Epidemiologic Studies Depression (CES-D) scale | Day 17
  The Center for Epidemiologic Studies Depression (CES-D) scale is a 20-item self-report measure of depressive symptoms. The range of scores is from 0 to 60, with higher scores reflecting increased depressive symptoms 41. The CES-D does not heavily depend on pathological items compared with other scales such as the Beck Depression Inventory and does not define clinical depression.
Positive and Negative Affect Schedule (PANAS ) | Day 17
  Positive and Negative Affect Schedule (PANAS ) is a 20-item scale that assesses both negative and positive affective states 44. Subjects rate adjectives describing affective states on a scale of 1 to 5 using a specified time period (e.g., now, today, past week etc.). Scores are then added up to generate negative and positive scale scores.
The Profile of Mood States (POMS) | Day 17
  The Profile of Mood States (POMS) is a 72-item questionnaire which consists of adjectives commonly used to describe momentary mood states. It has been found to be sensitive to the mood-altering effects of drugs including nicotine. POMS has a 5-point objective rating scale (0=not at all to 5=extremely). There are eight mood states that this scale measures: (1) Anger, (2) Anxiety, (3) Confusion, (4) Depression, (5) Elation, (6) Fatigue, (7) Friendliness and (8) Vigor. POMS will be used during each session to measure effects of atomoxetine or nicotine on mood.
Symptom Checklist Form (SCF) | Day 5
  In order to monitor adverse events from the study medications, SCF will be administered before and after each session. SCF is a locally developed symptom checklist that includes possible side effects of study medications with each symptom being scored 1-5.
Symptom Checklist Form (SCF) | Day 17
  In order to monitor adverse events from the study medications, SCF will be administered before and after each session. SCF is a locally developed symptom checklist that includes possible side effects of study medications with each symptom being scored 1-5.
Nicotine Withdrawal Symptom Checklist (NWSC) | Day 5
  Smokers will be asked to rate several nicotine withdrawal symptoms on a likert scale visual analogue. There are 12 items responses range from 0, "not at all" to 3 "extremely".
Nicotine Withdrawal Symptom Checklist (NWSC) | Day 17
  Smokers will be asked to rate several nicotine withdrawal symptoms on a likert scale visual analogue. There are 12 items responses range from 0, "not at all" to 3 "extremely".

CONTACTS AND LOCATIONS:
Overall Officials: Albert Arias, MD, Principal Investigator — Yale University
Locations (1):
- West Haven Veterans Affairs, West Haven, Connecticut, United States